CLINICAL TRIAL: NCT02869360
Title: Pilot Study of Positron Emission Tomography (PET) Imaging: Correlations With Advanced Magnetic Resonance Imaging in Multiple Sclerosis
Brief Title: Correlation Between PET and Advanced MRI in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Philippe Beauchemin, Clinical Fellow, University of British Columbia
Other Study IDs: CNS-2016-293
Record Dates: First submitted 2016-08-12; First posted 2016-08-16 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Multiple Sclerosis (MS) patients: 4 Secondary Progressive MS patients on no disease modifying therapy 4 Primary Progressive MS patients on no disease modifying therapy 4 Relapsing-Remitting MS patients on no disease modifying therapy 4 Relapsing-Remitting MS patients on Glatiramer Acetate 40 mg three times a week
- Healthy Controls: 4 Healthy volunteers aged between 18-60 years of age

SUMMARY:
Traditional Magnetic Resonance Imaging (MRI) in Multiple Sclerosis (MS) has enabled clinicians to measure disease activity but there are inherent limitations. Clinical/radiographic dissociation can be seen in some patients and the abnormalities are not specific.

This pilot study is an opportunity to determine the relationship between quantitative advanced MRI measures and OCT with PET measurements of microglial activation and myelin health.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Multiple Sclerosis according to the 2011 McDonald criteria.
* Aged 18 to 60
* High or mixed affinity binder to rs6971 TSPO polymorphism

Exclusion Criteria:

* Pregnant or breastfeeding
* Suffering from an unstable medical condition
* Have a neurological or ocular disorder other than MS
* Any contra-indications to MRI

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 4 untreated RRMS, 4 untreated SPMS, 4 untreated PPMS patients, 4 healthy controls and 4 GA 40mg TIW
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-10; Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Whole Brain PBR28 binding | Baseline

SECONDARY OUTCOMES:
Lesional PiB binding | Baseline
Myelin Water Imaging | Baseline
MR Spectroscopy (Total NAA, NAA/Cr, mI) | Baseline
Optical Coherence Tomography (RNFL thickness) | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- MS Clinical Trials Group - UBC, Vancouver, British Columbia, Canada